CLINICAL TRIAL: NCT05254236
Title: A Phase IIb, Randomized, Double-Blinded Trial to Evaluate the Immunogenicity and Safety Study of the Booster Dose Using the High or Medium Dose of COVID- 19 Vaccine (Vero Cell), Inactivated in Healthy Adults Who Have Completed Two Doses of mRNA Vaccine in Hong Kong
Brief Title: Immunogenicity and Safety Study of the 3rd Booster Dose Using the High or Medium Dose of Inactivated Vaccine in Healthy Adults in in Hong Kong
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Limited subjects
Sponsor: Sinovac Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO-nCOV-2004
Record Dates: First submitted 2022-02-20; First posted 2022-02-24 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medium-dose arm (Experimental): 75 participants vaccinated two doses of mRNA vaccine(prior to this study) will be given one dose booster immunization using medium-dose COVID-19 Vaccine (Vero Cell), Inactivated
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated (Medium-dose)
- High-dose arm (Experimental): 75 participants vaccinated two doses of mRNA vaccine(prior to this study) will be given one dose booster immunization using high-dose COVID-19 Vaccine (Vero Cell), Inactivated
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated (High-dose)

INTERVENTIONS:
Biological: COVID-19 Vaccine (Vero Cell), Inactivated (Medium-dose) — Medium-dose COVID-19 Vaccine(Vero Cell),Inactivated: 600SU inactivated SARS-CoV-2 virus in 0.5 mL of aluminium hydroxide solution per injection
  Other Names: Medium-dose CoronaVac®
  Arms: Medium-dose arm
Biological: COVID-19 Vaccine (Vero Cell), Inactivated (High-dose) — High-dose COVID-19 Vaccine(Vero Cell),Inactivated:1200SU inactivated SARS-CoV-2 virus in 0.5 mL of aluminium hydroxide solution per injection
  Arms: High-dose arm

SUMMARY:
This is a randomized, double-blinded, Phase IIb clinical trial of COVID-19 vaccine (CoronaVac®) manufactured by Sinovac Research & Development Co., Ltd.The purpose of this study is to evaluate to evaluate the changes in immunogenicity before and after the booster vaccine using the high (1200 SU) or medium (600 SU) dose of COVID-19 Vaccine (Vero Cell), Inactivated.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, Phase IIb clinical trial of 150 participants aged 18 years and above, who have completed two doses of mRNA COVID-19 vaccine as the primary vaccination for at least six months after the second dose. After enrollment, participants will be randomly assigned into two study arms at a ratio of 1:1 to receive a booster of one dose of medium-dose (600 SU) or one dose of high-dose (1200 SU) COVID-19 Vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 years and above, who have received two prior doses of mRNA COVID-19 vaccine (Comirnaty®, made by BioNTech/Pfizer) as the primary vaccination, with the second dose given at least 180 days prior to the day of booster vaccination in the present study;
* Evidence of a deep throat saliva (DTS) PCR negative for SARS-COV-2 within 24 hours before enrollment;
* Female participants who have a negative pregnancy test on the day of vaccination, and not currently breastfeeding;
* The participants are able to understand and sign the informed consent voluntarily;
* The participants are willing and able to comply with all schedule visits, sample collection,vaccine plan, and other study procedures;
* The participants must be willing to provide verifiable identification (in accordance with the local regulations), has means to be contacted and to contact the investigator during the study.

Exclusion Criteria:

* History of confirmed or having evidence showing a current infection of SARS-CoV-2 prior to randomization;
* Any prior administration of another investigational coronavirus vaccine or current/planned simultaneous participation in another interventional study to prevent or treat COVID-19;
* Known allergy to vaccines or vaccine ingredients, and serious adverse reactions to vaccines, such as urticaria, dyspnea, angioneurotic edema;
* Serious chronic disease, serious cardiovascular disease, hypertension and diabetes that cannot be controlled by drugs, hepatorenal disease, malignant tumor, etc.;
* Acute central nervous system diseases such as encephalitis/myelitis, acute disseminating encephalomyelitis, and related disorders;
* Receipt of blood/plasma products or immunoglobulins in the past three months before vaccination in this study;
* Participation in other studies involving study intervention within 30 days prior to vaccination in this study;
* Receipt of attenuated live vaccines in the past fourteen days prior to vaccination in this study;
* Receipt of inactivated or subunit vaccines in the past seven days prior to vaccination in this study;
* Acute exacerbation or presentation of stable chronic diseases (including but not limited to asthma,migraine, gastrointestinal disorder, etc.);
* Acute febrile illness with oral temperature >37.5C on the day of vaccination;
* According to the investigator's judgment, the participant has any other factors that might interfere with the results of the clinical trial or pose additional risk to the participant due to participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity index-Geometric mean fold rise (GMFR) of neutralization antibody titre in the high dose | 28 days after the booster dose vaccination
  Geometric mean fold rise (GMFR) of neutralization antibody titre from baseline to 28 days post the booster vaccine in the high dose .
Immunogenicity index-Geometric mean fold rise (GMFR) of neutralization antibody titre in the medium dose | 28 days after the booster dose vaccination
  Geometric mean fold rise (GMFR) of neutralization antibody titre from baseline to 28 days post the booster vaccine in the medium dose .

SECONDARY OUTCOMES:
Immunogenicity index-the seropositivity rate of neutralizing antibody in the high dose | 28 days after the booster dose vaccination
  The seropositivity rate of neutralizing antibody on day 28 after the booster dose vaccination in the high dose
Immunogenicity index-the seropositivity rate of neutralizing antibody in the medium dose | 28 days after the booster dose vaccination
  The seropositivity rate of neutralizing antibody on day 28 after the booster dose vaccination in the high dose
Immunogenicity index-Geometric mean of neutralizing antibody titer (GMT) in the medium dose | 28 days after the booster dose vaccination
  Geometric mean of neutralizing antibody titer (GMT) on Day 28 after the booster dose vaccination in the high dose
Immunogenicity index-Geometric mean of neutralizing antibody titer (GMT)in the medium dose | 28 days after the booster dose vaccination
  Geometric mean of neutralizing antibody titer (GMT) on Day 28 after the booster dose vaccination in the medium dose
Immunogenicity index-The seropositivity rate of neutralizing antibody in the high dose | 3 months after the booster dose vaccination
  The seropositivity rate of neutralizing antibody at 3 months after the booster dose vaccination in the high dose
Immunogenicity index-The seropositivity rate of neutralizing antibody in the medium dose | 3 months after the booster dose vaccination
  The seropositivity rate of neutralizing antibody at 3 months after the booster dose vaccination in the medium dose
Immunogenicity index-The seropositivity rate in the high dose | 6 months after the booster dose vaccination
  The seropositivity rate of neutralizing antibody at 6 months after the booster dose vaccination in the high dose
Immunogenicity index-The seropositivity rate in the medium dose | 6 months after the booster dose vaccination
  The seropositivity rate of neutralizing antibody at 6 months after the booster dose vaccination in the medium dose
Immunogenicity index-GMT of neutralizing antibody in the high dose | 3 months after the booster dose vaccination
  GMT of neutralizing antibody at 3 months after the booster dose vaccination in the medium dose
Immunogenicity index-the GMT of neutralizing antibody in the high dose | 6 months after the booster dose vaccination
  GMT of neutralizing antibody at 6 months after the booster dose vaccination in the medium dose
Immunogenicity index-GMT of neutralizing antibody in the medium dose | 3 months after the booster dose vaccination
  GMT of neutralizing antibody at 3 months after the booster dose vaccination in the medium dose
Immunogenicity index-the GMT of neutralizing antibody in the medium dose | 6 months after the booster dose vaccination
  GMT of neutralizing antibody at 6 months after the booster dose vaccination in the medium dose
Safety index-Occurrence, intensity, duration, and relationship of solicited local and systemic AEs | 28 days after the booster dose vaccination
  Occurrence, intensity, duration, and relationship of solicited local and systemic AEs for seven days following the booster dose vaccination and of unsolicited AEs for 28 days post booster vaccination.
Safety index-Occurrence and relationship of SAEs | Within 12 months post booster vaccination
  Occurrence and relationship of SAEs within 12 months post booster vaccination.
Safety index-Occurrence and relationship of AESI | Within 12 months post booster vaccination
  Occurrence and relationship of AESI within 12 months post booster vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Fan Ngai HUNG, Doctor, Principal Investigator — Gleneagles Hospital HongKong
Locations (1):
- Gleneagles Hospital HongKong, Hong Kong, China